CLINICAL TRIAL: NCT05494450
Title: An Open, Non-comparative, Multicenter Investigation to Evaluate the Safety and Performance of Exufiber Ag+, a Gelling Fiber Silver Dressing, When Used in Medium to High Exuding Chronic Wounds
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision secondary to data collection
Sponsor: Molnlycke Health Care AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ExufiberAg+02
Record Dates: First submitted 2022-08-08; First posted 2022-08-10 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Pressure Ulcer; Diabetic Foot Ulcer; Venous Leg Ulcer
MeSH Terms: conditions — Pressure Ulcer; Diabetic Foot; Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- ExufiberAG+02 (Other): using ExufiberAG as the primary dressing on medium to high exuding chronic wounds.
  Interventions: Device: ExufiberAG+

INTERVENTIONS:
Device: ExufiberAG+ — confirm performance and safety of the Exufiber Ag+ dressing in medium to high exuding chronic wounds

SUMMARY:
An open, non-comparative, multicenter investigation to evaluate the safety and performance of Exufiber Ag+, a gelling fiber silver dressing, when used in medium to high exuding chronic wounds

DETAILED DESCRIPTION:
The overall objective of this post market clinical follow-up (PMCF) investigation is to confirm performance and safety of the Exufiber Ag+ dressing in medium to high exuding chronic wounds, with Mepilex Border Flex as the secondary dressing, when used in accordance with the Instructions for Use.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form
2. Patient aged ≥18 years old
3. Patient with moderate to high exuding chronic wound (PU (stage II-IV), VLU or DFU)
4. Patient with target wound that is a shallow to deep wound or cavity
5. Patient with target wound that is ≥ 4 weeks in age
6. Patient with target wound that is ≥ 8 cm2

Exclusion Criteria:

1. Patient is contraindicated for the dressing according to product labeling
2. Known allergy/hypersensitivity to any of the components of the investigation products
3. Pregnancy/lactating female
4. Patient with spreading soft tissue infection/cellulitis in the wound (as judged by the Investigator)
5. Patient with known immunodeficiency
6. Patient taking systemic antibiotics
7. Patient with the target wound located on an infected limb and/or interfered by minimal blood flow in the opinion of the Investigator.
8. Patient with the target wound with an unexplored enteric fistula
9. Patient requiring treatment with oxidizing agents such as hypochlorite solutions or hydrogen peroxide
10. Patient who, in the opinion of the Investigator, is not expected to comply with the investigation due to physical and/or mental conditions
11. Patient who was previously enrolled in this investigation
12. Patient participating in other investigations that would preclude the subject from participating in this investigation as judged by the Investigator
13. Patient involved in the planning and conduct of the clinical investigation (applies to all Mölnlycke staff, investigational site staff, and third party vendor)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-11-29 (Actual); Study Completion 2022-11-29 (Actual)

PRIMARY OUTCOMES:
evaluate the safety and performance of Exufiber Ag+ in medium to high exuding chronic wounds | 28 Days
  open, non-comparative, multicenter investigation

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Center for Clinical Research, San Francisco, California
  - Sycamore Wound Care and Hyperbaric Center, Miamisburg, Ohio

IPD SHARING:
Plan to Share IPD: No